CLINICAL TRIAL: NCT05716360
Title: Early Postprocedural Susceptibility-Weighted Imaging and Vessel-Wall Imaging For Prediction of Complications After Flow-Diversion Treatment of Intracranial Aneurysms
Brief Title: Early Postprocedural Susceptibility-Weighted Imaging and Vessel-Wall Imaging For Prediction of Complications After Flow-Diversion Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Rifat Ozpar, Assistant Professor, Uludag University
Other Study IDs: TSG-2022-914
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Early Susceptibility-Weighted Imaging and Vessel-Wall Imaging Findings After Flow-Diversion Treatment of Intracranial Aneurysms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Aneuryms treated with Flow-Diverting Stents and had a diameter above 8 mm
  Interventions: Diagnostic Test: Pre-procedural, early and late post-procedural susceptibility weighted imaging and vessel wall imaging with a 3T Magnetic Resonance Imaging Device; Procedure: Aneurysm Treatment with Flow-Diversion Therapy
- Group 2: Aneuryms treated with Flow-Diverting Stents and had a diameter below 8 mm
  Interventions: Diagnostic Test: Pre-procedural, early and late post-procedural susceptibility weighted imaging and vessel wall imaging with a 3T Magnetic Resonance Imaging Device; Procedure: Aneurysm Treatment with Flow-Diversion Therapy
- Group 3: Aneurysms treated with metalic bare stents
  Interventions: Diagnostic Test: Pre-procedural, early and late post-procedural susceptibility weighted imaging and vessel wall imaging with a 3T Magnetic Resonance Imaging Device; Procedure: Aneurysm Treatment with Metalic Bare Stent

INTERVENTIONS:
Diagnostic Test: Pre-procedural, early and late post-procedural susceptibility weighted imaging and vessel wall imaging with a 3T Magnetic Resonance Imaging Device — Pre-procedural, early and late post-procedural susceptibility weighted imaging and vessel wall imaging with a 3T Magnetic Resonance Imaging Device
Procedure: Aneurysm Treatment with Flow-Diversion Therapy — Aneurysm Treatment with Flow-Diversion Therapy
  Groups: Group 1; Group 2
Procedure: Aneurysm Treatment with Metalic Bare Stent — Aneurysm Treatment with Metalic Bare Stent
  Groups: Group 3

SUMMARY:
Purpose: Examination of microangiopathic changes that may develop after flow-directed stenting of intracranial aneurysms with susceptibility-weighted imaging (SWI), and vessel wall imaging (VWI) of vessel wall inflammation that may be associated with stenosis in the stented vessel and rupture of the aneurysm.

Methods: SWI and VWI examinations will be performed before and after treatment in patients who are planned for flow-directing aneurysm treatment. Clinical follow-up of the cases will be performed during the first 3 months post-procedure. At the end of the 3rd month, SAG and DDG findings related to and unrelated to intracranial hemorrhage will be detected by control imaging.

DETAILED DESCRIPTION:
Susceptibility-weighted imaging (SWI) and vessel wall imaging (VWI) are among the most recent magnetic resonance (MR) techniques used to evaluate the cerebral vascular system (1,2). SWI; In addition to detecting the damage caused by many cerebrovascular pathologies at the microvascular level more sensitively than other imaging methods, it is the only MR sequence that can be used to differentiate blood-iron-calcification. It is the most sensitive MR sequence for iron accumulation and calcification. In addition to cerebrovascular diseases, it can be used in neurodegenerative diseases, especially parkinsonism, in the evaluation of tumoral - infective processes that can go with calcification (3). Similarly, VWI; It is used with increasing frequency in current practice in the diagnosis of pathologies affecting the vessel wall such as dissection, atherosclerotic change, inflammation and vasculitic involvement that cannot be clearly distinguished by normal vessel imaging methods (4). For both SWI and VWI, an MR device infrastructure with at least 3T magnetic field strength is required (2,5). Both techniques have limited diagnostic capabilities at magnetic field strengths up to 1.5T.

In studies conducted with VWI, it is stated that staining detected with VWI on the aneurysm wall may have predictive properties in terms of rupture (6,7). In addition, microhemorrhages detected by SWI imaging have been reported to transform into large parenchymal hemorrhages due to perfusion changes (8). Distant bleeding occurs due to perfusion change in some of the aneurysm cases that receive flow-directing therapy (9). In addition, rupture of the aneurysm may occur in some of the cases in which this treatment is applied, and stent stenocclusion may occur in some (10-11).

In the light of the above information, we aimed to evaluate the relationship between microhemorrhages, which may be a precursor of large parenchymal hemorrhages, staining of the aneurysm wall that may reflect the potential for rupture with VWI, and vessel wall staining or hematoma, which may reflect the risk of stenocclusion, with SWI examination to be performed on a 3T MR device in cases of intracranial aneurysms that were treated with flow-guided therapy, and complications developing after treatment.

References:

1. Haacke EM, Mittal S, Wu Z, Neelavalli J, Cheng YC. Susceptibility-weighted imaging: technical aspects and clinical applications, part 1. AJNR Am J Neuroradiol. 2009 Jan;30(1):19-30.
2. Mandell DM, Mossa-Basha M, Qiao Y, et al. Vessel Wall Imaging Study Group of the American Society of Neuroradiology. Intracranial Vessel Wall MRI: Principles and Expert Consensus Recommendations of the American Society of Neuroradiology. AJNR Am J Neuroradiol. 2017 Feb;38(2):218-229.
3. Mittal S, Wu Z, Neelavalli J, Haacke EM. Susceptibility-weighted imaging: technical aspects and clinical applications, part 2. AJNR Am J Neuroradiol. 2009 Feb;30(2):232-52.
4. Lindenholz A, van der Kolk AG, Zwanenburg JJM, Hendrikse J. The Use and Pitfalls of Intracranial Vessel Wall Imaging: How We Do It. radiology. 2018 Jan;286(1):12-28.
5. Nam Y, Gho SM, Kim DH, Kim EY, Lee J. Imaging of nigrosome 1 in substantia nigra at 3T using multiecho susceptibility map-weighted imaging (SMWI). J Magn Reson Imaging. 2017;46:528-536.
6. Texakalidis P, Hilditch CA, Lehman V, Lanzino G, Pereira VM, Brinjikji W. Vessel Wall Imaging of Intracranial Aneurysms: Systematic Review and Meta-analysis. World Neurosurg. 2018 Sep;117:453-458.e1.
7. Santarosa C, Cord B, Koo A, Bhogal P, Malhotra A, Payabvash S, Minja FJ, Matouk CC. Vessel wall magnetic resonance imaging in intracranial aneurysms: Principles and emerging clinical applications. Interv Neuroradiol. 2020 Apr;26(2):135-146.
8. Lau KK, Wong YK, Teo KC, et al. Long-Term Prognostic Implications of Cerebral Microbleeds in Chinese Patients With Ischemic Stroke. J Am Heart Assoc. 2017 Dec 7;6(12):e007360.
9. Zhou G, Su M, Yin YL, Li MH. Complications associated with the use of flow-diverting devices for cerebral aneurysms: a systematic review and meta-analysis. Neurosurg Focus. 2017 Jun;42(6):E17.
10. Darsaut TE, Rayner-Hartley E, Makoyeva A, Salazkin I, Berthelet F, Raymond J. Aneurysm rupture after endovascular flow diversion: the possible role of persistent flows through the transition zone associated with device deformation. Interv Neuroradiol. 2013 Jun;19(2):180-5.
11. Klisch J, Turk A, Turner R, Woo HH, Fiorella D. Very late thrombosis of flow-diverting constructs after the treatment of large fusiform posterior circulation aneurysms. AJNR Am J Neuroradiol. 2011 Apr;32(4):627-32.

Study Protocol, Methods and Procedures:

Patients who are scheduled for endovascular treatment with a stent for their intracranial aneurysm following upgrading of the MR device will be included in the study. Cases will be divided into 3 groups according to the characteristics of aneurysms in digital subtraction angiography (DSA) examination. In Group 1, patients with a diameter greater than 8 mm and suitable for flow-guiding therapy, in Group 2. Patients with a diameter of less than 8 mm and suitable for flow-guiding therapy, in Group 3. Patients whose aneurysm is suitable for treatment with a metal-coated stent. will take. A total of 60 patients, 20 patients in each group, will be included in the study. Verbal and written informed consent will be obtained from all patients for imaging and treatments.

Patients to be included in the study will be examined in the last 24 hours prior to endovascular treatment in an elevated 3T MR device (preprocedural examination). SWI, VWI sequences will be obtained. In addition, the current neurological findings of the patients will be recorded. Control SWI and VWI sequences will be available within 48 hours of performing endovascular therapy (early postprocedural examination). In the preprocedural and postprocedural examinations, microbleeding foci detected in SWI and vessel wall inflammation findings observed in VWI will be recorded. Following the imaging, the clinic of the patients will be evaluated verbally on the 3rd day, 1st week, 1st month, 2nd month and 3rd month after treatment. In the 3rd month, the patient's neurological examination will be repeated and control SWI - VWI examinations will be performed (late postprocedural examination). Clinical symptoms that develop in the event of neurological deterioration will be recorded and the patient will be examined by cranial MR, cranial MR angiography and cranial computed tomography for intracranial bleeding, aneurysm rupture and stent occlusion. Cases out of follow-up will be excluded from the study.

In all 3 groups, the possible relationship between microhemorrhage foci in preprocedural, early and late postprocedural SWI and vessel wall inflammation findings in VWI and radiological findings such as bleeding or ischemia that may be related to worsening, worsening of clinical condition, various statistical findings, especially chi-square test. methods will be investigated. It will be evaluated whether the findings observed in SWI and VWI are predictive in terms of intracranial hemorrhage, aneurysm rupture and stent occlusion in patients who received current converter therapy. Findings that do not cause clinical symptoms and are observed in SWI and VWI will be determined in current converter cases. In addition, it will be investigated whether there is a significant difference between the SWI and VWI findings observed in the cases treated with current-converting treatment and those treated with metal-covered stent, and the possible effect of aneurysm size on SWI and VWI findings in cases treated with current-converting treatment.

ELIGIBILITY:
Inclusion Criteria:

Endovascular treatment plan with stent for intracranial aneurysm No kidney dysfunction history No MRI contrast material allergy history

Exclusion Criteria:

Pregnancy History of MR contrast material allergy Kidney dysfunction Leave Following-up During Study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are scheduled for endovascular treatment with a stent for their intracranial aneurysm following upgrading of the MR device will be included in the study. Cases will be divided into 3 groups according to the characteristics of aneurysms in digital subtraction angiography (DSA) examination. In Group 1, patients with a diameter greater than 8 mm and suitable for flow-guiding therapy, in Group 2. Patients with a diameter of less than 8 mm and suitable for flow-guiding therapy, in Group 3. Patients whose aneurysm is suitable for treatment with a metal-coated stent. will take. A total of 60 patients, 20 patients in each group, will be included in the study. Verbal and written informed consent will be obtained from all patients for imaging and treatments.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
Determining Clinical Significant and Unsignificant Early Post-procedural susceptibility weighted and vessel wall imaging findings related to flow diversion treatment of intracranial aneurysms | Post-procedural First Three Months

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University Faculty of Medicine Department of Radiology, Bursa, Nilufer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No